CLINICAL TRIAL: NCT01387048
Title: Phase IV An Evaluator-Blind Controlled Parallel-Group Study To Assess Efficacy And Safety Of Skinoren® 15% Gel And Differin® 0,1% Gel For The Treatment And Maintenance Treatment Of Facial Acne Vulgaris And Late-Type Acne In Females
Brief Title: Study for Long-term Treatment of Acne Vulgaris With Skinoren Versus Differin
Acronym: SKADI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Antje Wiede, Dr. rer. nat., University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BS-HAU-2011; 2011-000152-42 (EudraCT Number)
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; late-type acne; Skinoren; maintenance
MeSH Terms: conditions — Acne Vulgaris | interventions — azelaic acid; Adapalene; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Skinoren gel 15 %, topical (Experimental): primary treatment 12 weeks with Skinoren gel®, followed by maintenance therapy with Skinoren gel® for another 24 weeks,
  Interventions: Drug: skinoren
- Differin Gel 0.1% (Active Comparator): primary 12 weeks therapy with Differin gel®, followed by maintenance therapy with Differin gel® for another 24 weeks.
  Interventions: Drug: differin
- Skinoren (Experimental): primary 12 weeks therapy with Skinoren gel®, followed by observation only for another 24 weeks,
  Interventions: Drug: skinoren

INTERVENTIONS:
Drug: skinoren — gel 15%, twice daily, 36 weeks
  Other Names: Generikum
  Arms: Skinoren gel 15 %, topical
Drug: differin — 0.1% gel, once daily in the evening
  Other Names: Epiduo
  Arms: Differin Gel 0.1%
Drug: skinoren — 12 weeks treatment, the following 24 months only observation
  Other Names: Generikum
  Arms: Skinoren

SUMMARY:
The purpose of this study is to assess the effect of Skinoren® 15% gel compared to no therapy on the maintenance of clinical therapy success in subjects with mild to moderate acne vulgaris previously treated for 3 months by a monotherapy of this substance and to assess the effect of Skinoren® 15% gel, compared to Differin® 0.1% gel on the efficacy and safety during a 9-month long-term treatment period.

DETAILED DESCRIPTION:
Differin gel, containing adapalene 0.1%, has been used now for several years in the topical treatment of mild to moderate acne. It has comedolytic and anti-inflammatory activities,and is equally effective and less irritant than other topical retinoids. Adapalene has been shown to maintain therapeutic effect achieved after three months of monotherapy for further three months. Furthermore, its effect in maintenance therapy has been shown in several studies after initial combination with topical or systemic antimicrobials. Skinoren 15% gel (azelaic acid) is an alternative treatment affecting several pathogenetic factors of acne, which has potential in maintenance therapy due to its good tolerability and safety and missing contraindications concerning long-term treatment, which allow even use in pregnancy.

Azelaic acid (AzA; HOOC-(CH2)7-COOH) is a naturally occurring compound that interferes with acne pathogenesis by virtue of its antikeratinizing, antibacterial, and anti-inflammatory properties. Vehicle-controlled studies have verified that AzA exercises a significant and clinically relevant effect on both non-inflammatory and inflammatory acne lesions. In the treatment of moderate to severe acne, 20 percent AzA cream may be favorably combined with minocycline (90 percent good and excellent results), and may contribute towards reducing recurrences following discontinuation of systemic therapy (maintenance therapy with AzA cream). Particular advantages of AzA therapy include its favorable safety and side effect profile. It is non-teratogenic, is not associated with systemic adverse events or photodynamic reactions, exhibits excellent local tolerability, and does not induce resistance in Propionibacterium acnes. The 15 % azelaic acid gel has recently proven efficacy in a maintenance treatment of papulopustular rosacea after a combination treatment with oral doxycycline.

Mild to moderate acne vulgaris is defined as global severity of 2 through 4, according to the Investigator´s Static Global Assessment (ISGA) and Leeds Revised Acne Grading Scale from 2 trough 7.This inclusion criterion corresponds to the clinical grades usually treated with topical anti-acne therapies.

The non-treatment group during the maintenance phase helps to demonstrate the efficacy of Skinoren 15% gel in a maintenance treatment, thereby corroborating the necessity for maintenance therapy reflecting acne as a chronic disease.

Acne lesion counting has been used widely in the evaluation of new acne treatments as a change in facial acne lesions counts over time in an individual patient could reflect a true change. However, lesion counts are more valid in greater patient populations as planned in this study. Therefore, the lesion counts are defined as secondary efficacy criteria except during the maintenance phase for the population treated with azelaic acid. As described before, microcomedones are considered as precursor lesion. Moreover, their counts are constantly reduced during acne treatment and precede the clinical relapse. Therefore, microcomedones counts will be used in this trial as a marker of maintenance of therapeutic effect achieved during initial treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects between 18 and 45 years of age, inclusive, in good general health.
2. Female Subjects of childbearing potential using effective contraceptional methods must have been taking the same type of birth control for at least 6 months prior to entering the study and must not change type of birth control during the study. The subject´s should be willing to perform UPT in decision by physician, if indicated.
3. Subjects with mild to moderate acne vulgaris or late-type acne with global facial severity grade 2 through 4 according to the "Investigator´s Static Global Assessment (ISGA)" and B-G (2-7) according to the "Leeds revised acne grading system".
4. Subjects with visible microcomedones on the Cyanoacrylate strip taken on the forehead.
5. Subjects must read and sign the approved Informed Consent Form (and any local or national authorized requirements )prior to any participation in the study. Subjects must be willing and capable of cooperating to the extent and degree required by the protocol (including refraining from the use of cosmetics and ointments during the course of treatment). Subject must be able to follow all study procedures, attend all schedule visits, and complete the study successfully.

Exclusion Criteria:

1. Female subjects who are pregnant, trying to become or willing to become pregnant, or who are lactating.
2. Subjects who have any clinically relevant finding at their screening physical examination or medical history such as severe systemic diseases or diseases of the facial skin other than acne vulgaris (eg, acne conglobata, acne fulminans, secondary-acne or severe nodulocystic acne requiring treatment with oral isotretinoin).
3. Subjects who have a known hypersensitivity or previous allergic reaction to any of the active components of the study medication.
4. Subjects who are using and not willing to refrain from the following other types of facial products: astringents, toners, abradants, facials, peels containing glycolic or other acids, masks, washes or soaps.
5. Subjects who have used topical corticosteroids on the face or systemic corticosteroids within the past 2 weeks.
6. Subjects who have used topical antibiotics on the face or systemic antibiotics (only penicillin allowed) within the last 2 weeks.
7. Subjects who have used topical anti-acne medications within the past 2 weeks.
8. Subjects who have used systemic retinoids within the past 6 months.
9. Subjects who use medications that are reported to exacerbate acne
10. Subjects who are using drugs known to be photosensitizers because of the possibility of increased phototoxicity.
11. Subjects who have had a facial procedure performed by an esthetician, beautician, physician, nurse, or other practitioner, within the last 4 weeks.
12. Subjects who planned intensive UV exposure during study
13. Subjects who participated in another investigational drug or device research study within 30 days of enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Superiority of Skinoren 15% Gel | 36 weeks
  Superiority of Skinoren 15% Gel-group over the observational group in the maintanance phase. Change of Global Severity Grades (ISGA and Leeds)
Non-inferiority of Skinoren 15 % gel over the Differin 0.1% gel | 36 weeks
  Non-inferiority of Skinoren 15% Gel over the current "gold standard" Differin 0.1% gel in the long-term-treatment period: Change of Global severity grades

SECONDARY OUTCOMES:
- Change of non-inflammatory, inflammatory and total lesions at all visits. | 36 weeks
  - Secondary Endpoints:
  Microcomedone count changes from week 12-36
Change of non-inflammatory, inflammatory and total lesions at all visits | 36 weeks
  Subjects efficacy assessment
change of non-inflammatory, inflammatory and total lesions at all visits | 36 weeks
  subjects tolerability assessment
Change of non-inflammatory, inflammatory and total lesions at all visits | 36 weeks
  Subjects DLQI assessment
change of non-inflammatory, inflammatory and total lesions at all visits | 36 weeks
  Investigators tolerability assessment
change of non-inflammatory, inflammatory and total lesions at all visits | 36 weeks
  Relapse rate: Number of subjects which lose more than 50% of their initial improvement achieved at maintanance phase

CONTACTS AND LOCATIONS:
Overall Officials: Anja Thielitz, Dr. med., Principal Investigator — unfillated
Locations (1):
- Clinic for Dermatology and Vereology, Central Hospital Magdeburg, Magdeburg, Saxony-Anhalt, Germany